CLINICAL TRIAL: NCT03580759
Title: A Home-based Pre-Surgical Exergaming Intervention for Individuals With Advanced HF and Multiple Chronic Conditions Prior to Left Ventricular Assist Device Implantation or Heart Transplant
Brief Title: Exergaming in Advanced HF With Multiple Chronic Conditions Prior to LVAD Implantation or Heart Transplant
Acronym: PREHAB-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0407-18-FB
Record Dates: First submitted 2018-06-13; First posted 2018-07-09 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Heart-Assist Devices; Heart Failure NYHA Class IV; Exercise Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergaming (Experimental): Subjects in the exergaming group will participate in three exergaming training sessions with the Wii Fit U exergaming system. The Wii Fit U will then be left in the subjects' homes for a minimum of four weeks prior to left ventricular assist device implantation or heart transplant.
  Interventions: Behavioral: PREHAB
- Usual Care (No Intervention): Subjects in the usual care group will be encouraged to partake in physical activity as recommended in the 2017 AHA/ACC/HFSA guidelines for heart failure.

INTERVENTIONS:
Behavioral: PREHAB — After three supervised training sessions, subjects will be asked to participate in a daily exergaming activity tailored to their physical activity capabilities and needs. Subjects will be taught to rate their perceived exertion and monitor their target heart rate using a Fit Bit Charge HR. Daily exercise diaries will be used to monitor subject-perceived progress throughout the intervention period.
  Arms: Exergaming

SUMMARY:
The purpose of this study is to test a home-based exergaming intervention designed to decrease frailty and fatigue and improve affective well-being, functional capacity, and immune function in individuals with advanced heart failure (HF) and multiple chronic conditions (MCC) prior to receiving either a left ventricular assist device (LVAD) or orthotopic heart transplantation (OHT). Prior to surgery, individuals with advanced HF/MCC experience a high symptom burden that often precludes them from participating in meaningful physical activity. Pre-surgical fitness programs have been used in other critically ill populations to improve function prior to surgery. Interactive gaming systems have been successfully used to engage other seriously ill adults in low-intensity physical activity. However, exergaming interventions have not yet been applied in individuals with advanced HF/MCC as prehabilitation prior to LVAD implantation or OHT. The investigators propose that a prehabilitation exergaming intervention will not only enhance pre-surgical outcomes but will also augment postoperative outcomes. This study is designed in two-phases. Phase 1 examines intervention feasibility and phase 2 is a pilot study with a two-group design. In phase 2, participants will be randomized to a usual care group or the exergaming intervention group. The exergaming group will participate in a low-intensity exergaming intervention and additional investigator-developed educational modules that will be delivered via the Nintendo Wii U exergaming system. The investigators will evaluate pre- and post-surgical frailty, fatigue, affective well-being, and immune function as primary outcomes. The investigators expect that participation in low intensity exergaming will improve these primary outcomes pre- and post-surgically, and decrease post-surgical complications and health care utilization. Investigator-developed modules will promote self-efficacy, self-regulation, and activation. This is the first study to apply low-intensity exergaming to a pre-operative advanced HF/MCC population. The successful application of this intervention has significant implications to the pre-operative conditioning of individuals with advanced HF/MCC prior to LVAD implantation or OHT.

DETAILED DESCRIPTION:
Specific Aims. The objectives of this study are two-fold: (1) To test the feasibility of a low intensity, home-based exergaming intervention in individuals with advanced HF/MCC prior to left ventricular assist device (LVAD) implantation or orthotopic heart transplantation (OHT), and (2) To examine the effectiveness of delivering a low intensity, home-based exergaming intervention to decrease frailty and fatigue and improve affective well-being, functional capacity, and immune function in individuals with advanced HF/MCC prior to receiving an LVAD or OHT.

Other surgical populations who were deconditioned, fatigued, and frail before surgery have benefited from the use of pre-surgical fitness interventions (prehabilitation).3-5 Innovative interventions strategies, like the Nintendo Wii Fit exergaming system, have been successful at engaging seriously ill adults in low-intensity physical activity6,7. However, exergaming interventions have not yet been applied in individuals with advanced HF as prehabilitation prior to LVAD implantation or OHT. The investigators propose that a home-based, prehabilitation exergaming intervention will not only enhance pre-surgical outcomes but will also augment postoperative outcomes.

The investigators will conduct this study in two phases. Phase 1 is designed as a feasibility study in a smaller sample (5 participants and 5 informal caregivers) to allow initial evaluation of the intervention including troubleshooting the technological components and evaluating study recruitment, retention, and intervention safety prior to initiating the larger, two-group randomized study. Phase 2 will enroll a convenience sample of 40 participants with advanced HF/MCC who are being evaluated for LVAD implantation or OHT at Nebraska Medicine and their 40 informal caregivers for a total sample of 80 enrollees (n=40 exergaming, n=40 usual care).

In both phases, the exergaming group will participate in a low-intensity exergaming intervention and additional investigator-developed educational modules (e.g. symptoms while exercising, exercising with heart failure) that will be delivered via the Nintendo Wii U exergaming system. Investigator-developed modules are designed to promote self-efficacy, self-regulation, and activation. Individuals with advanced HF/MCC will be expected to participate in the exergaming intervention and the investigator-developed modules. Caregivers will be asked to be present for all training sessions and participate in the investigator-developed modules. The investigators will evaluate pre- and post-surgical frailty, fatigue, affective well-being, and immune function as primary outcomes in the individuals with advanced HF/MCC. The investigators expect that participation in low intensity exergaming will improve these primary outcomes pre- and post-surgically, and decrease post-surgical complications and health care utilization. Relationships will be examined among self-efficacy, self-regulation, and activation scores over time, and adherence to the intervention to test whether self-management mechanisms were effective in promoting adherence. Additionally, post-intervention qualitative interviews will be conducted to assess participant and caregiver experiences with the intervention.

Specific aims of this study are the following:

Aim 1 (Phase 1): Evaluate the feasibility of the home-based, low intensity exergaming intervention in individuals with advanced HF/MCC prior to LVAD implantation or OHT and their informal caregivers by assessing recruitment, enrollment, acceptability, adherence, subjects perception of barriers and facilitators, and implementation (delivery, fidelity, and procedures for data collection).

Aim 2 (Phase 2): Evaluate the impact of home-based, low intensity exergaming on pre- and post-surgical outcomes: frailty, fatigue, affective well-being, immune function, and biomarkers of co-morbid conditions at baseline, 4 weeks, and 1 and 3 months post-surgery compared to usual care (All subjects with advanced HF/MCC).

H1. Subjects in the exergaming group will have decreased frailty and fatigue and improved affective well-being and immune function compared to usual care.

Aim 3 (Phase 2): Evaluate the impact of home-based, low intensity exergaming on post-surgical complications (death, infection, bleeding, and rejection) and health care utilization (emergency department visits, unplanned hospital admissions) compared to usual care (both groups of subjects).

H2.a. Subjects in the exergaming group will have fewer post-surgical complications compared to usual care.

H2.b. Subjects in the exergaming group will have fewer emergency department visits and hospital admissions compared to usual care.

Aim 4 (Phase 2): Explore relationships among self-efficacy, self-regulation, and activation scores over time, intervention adherence, and pre- and post-surgical outcomes (Exergaming group participants and caregivers only).

There is a critical need to address deconditioning, fatigue, and frailty in individuals with advanced HF/MCC prior to LVAD implantation or OHT. This innovative exergaming intervention incorporates the use of an interactive, home-based technology to improve pre-and post-surgical outcomes

ELIGIBILITY:
Inclusion Criteria for Participants:

* age >19 years
* diagnosis of advanced HF and a minimum of one additional co-occurring chronic condition
* undergoing evaluation for left ventricular assist device implantation or heart transplant
* medical clearance from a heart failure cardiologist in the Nebraska Medicine Advanced HF Clinic.
* the ability to speak and understand English

Inclusion Criteria for Caregivers:

* age>19 years
* the ability to speak and understand English

Exclusion Criteria for Participants:

* cognitive impairment (Montreal Objective Cognitive Assessment39 [MoCA] < 26), -neuromuscular or orthopedic impairment that would preclude low-intensity physical activity
* unwillingness to complete two supervised sessions in the clinical setting, and one in the home setting
* ongoing inotrope therapy. (Exercise is discouraged during inotrope therapy.)
* inability to pass a Wii Fit Balance Board safety screen (prior to randomization in Phase 2)

Exclusion criteria for Caregivers:

* Unwillingness to participate in the supervised exergaming training sessions
* Unwillingness to participate in final qualitative interview

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Functional Capacity from Baseline | Baseline, 1 month post-intervention, 1 & 3 months post-surgery
  Functional capacity will be assessed with a six-minute walk test. Subjects will be asked to walk for 6 min to determine what distance they can accomplish in that time period at a normal walking pace.
Change in Physical Frailty from Baseline | Baseline, 1 month post-intervention, 1 & 3 months post-surgery
  Physical frailty will be assessed using the Fried criteria which include: Unintentional weight loss (10 lbs in past year), exhaustion, weakness (grip strength), slow walking speed, and low physical activity (0 criteria-not frail; 1-2 criteria-pre-frail; ≥3-frail)
Change in Fatigue from Baseline | Baseline, 1 month post-intervention, 1 & 3 months post-surgery
  Fatigue will be assessed with the NINR Fatigue Common Data Element which is a 6-item self-report 5-item Likert scale. Higher scores indicate greater feelings of fatigue. Max score is 30.

SECONDARY OUTCOMES:
Change in Immune Function from Baseline | Baseline, 1 month post-intervention, 1 & 3 months post-surgery
  Immune function will be assessed with a cell-mediated immune function assay (ImmuKnow) that is commercially available.

CONTACTS AND LOCATIONS:
Overall Officials: Windy W Alonso, PhD, RN, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No